CLINICAL TRIAL: NCT02896491
Title: Radiofrequency Electromagnetic Fields (RF-EMF) Effects on Brain Activity During Wake and Sleep in Healthy Elderly Males
Brief Title: RF-EMF Effects on the CNS in Elderly Men
Acronym: EMF60+males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Federal Office for Radiation Protection, Germany (Other Government)
Collaborators: Seibersdorf Labor GmbH (Industry)
Responsible Party: Principal Investigator, Heidi Danker-Hopfe, Ph.D., Head of Competence Center of Sleep Medicine and Sleep Research, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 3616S82430
Record Dates: First submitted 2016-05-27; First posted 2016-09-12 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Non-Ionizing Radiation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSM 900 MHz exposure (Experimental): Radiation: Exposure with non-ionizing electromagnetic fields exposure with GSM 900 MHz (2W/kg)
  Interventions: Radiation: Exposure with non-ionizing electromagnetic fields
- TETRA 400 MHz exposure (Experimental): Radiation: Exposure with non-ionizing electromagnetic fields:
  exposure with TETRA (6W/kg)
  Interventions: Radiation: Exposure with non-ionizing electromagnetic fields
- Sham exposure (Sham Comparator): Radiation: Exposure with non-ionizing electromagnetic fields: exposure with 0 W/kg
  Interventions: Radiation: Exposure with non-ionizing electromagnetic fields

INTERVENTIONS:
Radiation: Exposure with non-ionizing electromagnetic fields — In a cross-over design subjects will be exposed to sham (placebo), GSM 900 MHz (2W/kg) and TETRA (6W/kg)

SUMMARY:
To investigate possible effects of radio frequency electromagnetic fields on EEG activity during sleep and on Brain function during wake (EEG in the resting state condition, slow EEG potentials, auditory evoked potentials) and cognitive performance measures in test of selective attention, divided attention and working memory in healthy elderly males (60 - 80 years).

DETAILED DESCRIPTION:
To investigate possible effects of radio frequency electromagnetic fields on EEG activity during sleep and on Brain function during wake (EEG in the resting state condition, slow EEG potentials, auditory evoked potentials) and cognitive performance measures in test of selective attention, divided attention and working memory in healthy elderly males (60 - 80 years).

Subjects will be exposed with signals from mobile communication handheld devices for 7.5 h during the night and for the whole duration of the test session during the day. Exposures will be GSM (900 MHz), TETRA (400 MHz) and sham. Each subject is exposed with each exposure three times in addition to an adaptation/screening night and day to learn the test.

The results have to be discussed in the context of possible health risks resulting from RF-EMF exposure.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects (age 60 - 80 years)
* right handedness
* alpha EEG as resting state EEG
* non-smokers

Exclusion Criteria:

* acute illness
* severe neurological, psychiatric or internal disease
* CNS active medication
* sleep disorders
* drug abuse

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-01; Primary Completion 2018-01-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
sleep EEG (power) | during exposure for 8 hours

SECONDARY OUTCOMES:
resting state Waking EEG (power) | during exposure 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Blanka Pophof, Ph.D, Study Chair — Federal Office of Radiation Protection
Locations (1):
- Competence Center Sleep Medicine, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eggert T, Dorn H, Sauter C, Schmid G, Danker-Hopfe H. RF-EMF exposure effects on sleep - Age doesn't matter in men! Environ Res. 2020 Dec;191:110173. doi: 10.1016/j.envres.2020.110173. Epub 2020 Sep 12. PMID 32931791
- [Derived] Danker-Hopfe H, Dorn H, Sauter C, Schmid G, Eggert T. An experimental study on effects of radiofrequency electromagnetic fields on sleep in healthy elderly males and females: Gender matters! Environ Res. 2020 Apr;183:109181. doi: 10.1016/j.envres.2020.109181. Epub 2020 Jan 24. PMID 32014649